CLINICAL TRIAL: NCT05395195
Title: Erythropoietin Monotherapy for Brain Regeneration in Neonatal Encephalopathy in Low and Middle-Income Countries
Brief Title: Erythropoietin for Neonatal Encephalopathy in LMIC (EMBRACE Trial)
Acronym: EMBRACE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5623613
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Encephalopathy; Erythropoietin; Newborn Asphyxia
MeSH Terms: conditions — Brain Diseases; Asphyxia Neonatorum | interventions — Erythropoietin

STUDY DESIGN:
Intervention Model Description: Erythropoietin (intravenous or subcutaneous)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All injections with be administered behind a screen by dedicated personnel. The control arm will have mock (pretend) injections.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Erythropoietin (Experimental): Intravenous or subcutaneous injections of erythropoietin (500 U/kg/dose). Total of 9 doses will be administered. First dose will be given within 6 hours of birth. Second dose between 12 to 24 hours from the first dose. Subsequent 7 doses every 24 hours from the second dose.
  Interventions: Drug: Erythropoietin; Other: Supportive neonatal intensive care
- Control (Sham Comparator): Mock administration of injections (pretend) behind a screen by a dedicated personal
  Interventions: Other: Supportive neonatal intensive care

INTERVENTIONS:
Drug: Erythropoietin — Erythropoietin injections (500u/kg) x 9 doses
  Arms: Erythropoietin
Other: Supportive neonatal intensive care — Neonatal intensive care monitoring and support including ventilatory and inotropic support as clinically indicated

SUMMARY:
One million babies die, and at least 2 million survive with lifelong disabilities following neonatal encephalopathy (NE) in low and middle-income countries (LMICs), every year. Cooling therapy in the context of modern tertiary intensive care improves outcome after NE in high-income countries. However, the uptake and applicability of cooling therapy in LMICs is poor, due to the lack of intensive care and transport facilities to initiate and administer the treatment within the six-hours window after birth as well as the absence of safety and efficacy data on hypothermia for moderate or severe NE.

Erythropoietin (Epo) is a promising neuroprotectant with both acute effects (anti-inflammatory, anti-excitotoxic, antioxidant, and antiapoptotic) and regenerative effects (neurogenesis, angiogenesis, and oligodendrogenesis),which are essential for the repair of injury and normal neurodevelopment when used as a mono therapy in pre-clinical models (i.e without adjunct hypothermia).

The preclinical data on combined use of Eythropoeitin and hypothermia is less convincing as the mechanisms overlap. Thus, the HEAL (High dose erythropoietin for asphyxia and encephalopathy) trial, a large phase III clinical trial involving 500 babies with with encephalopathy reported that that Erythropoietin along with hypothermia is not beneficial.

In contrast, the pooled data from 5 small randomized clinical trials (RCTs) (n=348 babies), suggests that Epo (without cooling therapy) reduce the risk of death or disability at 3 months or more after NE (Risk Ratio 0.62 (95% CI 0.40 to 0.98). Hence, a definitive trial (phase III) for rigorous evaluation of the safety and efficacy of Epo monotherapy in LMIC is now warranted.

DETAILED DESCRIPTION:
The burden of neonatal encephalopathy is far higher in low and middle-income countries. Recently, the Hypothermia for Encephalopathy in Low and Middle-Income Countries Trial (HELIX) study concluded cooling therapy did not reduce the combined outcome of death or disability at 18 months after neonatal encephalopathy in low-income and middle-income countries. In fact, the results found that cooling therapy significantly increased death alone. This warrants exploration of the efficacy of other treatment adjuncts for these settings.

One medication with potential for monotherapy is Erythropoietin. Erythropoietin is an erythropoiesis stimulating cytokine used for the treatment of anaemia. It is a Food and Drug Administration (FDA) approved drug that is widely used for treatment of anaemia including premature babies and has extensive safety profile in newborn babies.

Erythropoietin is also produced by neurons and glia in the hippocampus, internal capsule, cortex, and midbrain in response to hypoxia. More recently, erythropoietin has been reported as having anti-apoptotic, anti-inflammatory and anti-oxidative effects, making it a prime neuroprotective candidate. It also reduces free iron accumulation which occurs due to hypoxic ischemia by inducing erythropoiesis, which promotes neurogenesis. Extensive preclinical small and large animal models have demonstrated neuroprotective and neuro reparative effects of Erythropoietin when used as monotherapy.

A number of small randomised controlled trials have been reported from low and middle-income countries. A systematic review and meta-analysis of Erythropoietin monotherapy in babies with neonatal encephalopathy in LMIC showed pooled data including a total of 348 babies from 5 clinical trials in LMIC suggest 40% relative risk reduction (Risk Ratio 0.62 (95% Confidence Intervals (CI) 0.40 to 0.98) in death or disability at 18 months with Erythropoietin, compared with placebo. None of these clinical trials have reported any serious adverse events of Erythropoietin monotherapy.

Erythropoietin dose used in these trials varied from 300U/kg to 2500U/kg, single dose to a maximum of two weeks of duration starting within 24 hours after birth. The largest of these trials, reported from China have used a low dose (500U/kg) on alternate days for two weeks. This trial recruited 153 babies with moderate or severe encephalopathy and reported that Erythropoietin significantly reduced death or disability at 18 months.

More recently, another randomised controlled trial of Erythropoietin involving 62 normothermic babies with moderate or severe neonatal encephalopathy has been reported from Government Medical College, Aurangabad in India. The investigators used an Erythropoietin dose of 500 U/kg alternate days for 10 days starting within 24 hours. Neonatal mortality was significantly lower (39%; 12/31) in the Erythropoietin group compared with the placebo group (71%; 22/31) (p=0.01). No adverse events were reported in the Erythropoietin group.

The EMBRACE trial is a phase III, multi-country, double-blinded, placebo-controlled randomised controlled trial of Erythropoietin versus sham injection (placebo) in babies with neonatal encephalopathy in low and middle-income countries. All clinical and study team except for the nurse administering the trial drug will be masked to the intervention. The investigators plan to randomise 504 babies in this trial. The dosing regimen will be IV/Sub cutaneous Erythropoietin 500unit/kg within 6 hours of birth and then daily until 8 days. In total, there will be 9 doses. Body temperature of all babies will be monitored 4 hourly for the first three days after birth and normothermia (36.0-37.5°C) will be maintained as a part of the usual care at these hospitals with an algorithm to prevent/treat hyperthermia.

Magnetic resonance biomarkers including spectroscopy and diffusion tensor imaging will be acquired between 1 to 2 weeks of age in all recruited babies. The MR scanners and sequences at each site will be harmonised prior to recruitment.

The trial will have an 18 month recruitment period, a 18 month follow-up period, and 5 months for data analysis and write up. A pilot study (external pilot) of 50 babies will be done prior to the start of the EMBRACE trial (Jan 2023 to April 2023) but these patients will not be included in the main trial. Minor updates to the trial protocol may be made after the completion of the pilot trial.

ELIGIBILITY:
Inclusion Criteria (all of below should be met)

* Inborn babies born at a gestational age greater than or equal to 36 weeks, with a birth weight >=1.8 kg
* At least one of the following: need for continued resuscitation at 5 minutes of age; 5-minute Apgar score < 6; metabolic acidosis (pH < 7.0; base deficit > 16 mmol/L) in cord or blood gas within the first hour of birth.
* Moderate or severe neonatal encephalopathy on modified Sarnat staging performed between 1 to 6 hours after birth.

Exclusion Criteria:

* Imminent death at the time of recruitment
* Babies born at home or those admitted after 6 hours of birth.
* Major life-threatening congenital malformations
* Head circumference <30 cm at birth
* Babies undergoing induced hypothermia
* Migrant family or parents unable/unlikely to come back for follow-up at 18 months
* Sentinel event and encephalopathy occurred only after birth
* Unable to consent in primary language of parent(s)

Ages: 1 Hour to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 504 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of babies who die or survive with moderate or severe disability | 18 to 22 months
  Death or moderate or severe disability in survivors

SECONDARY OUTCOMES:
Number of babies who die | Upto 22 months
  Mortality from all causes
Number of babies who survive without neurodisability | 18 to 22 months
  Survival with Bayley composite scale scores >84 in all domains, no cerebral palsy, no seizure disorder, hearing or visual defect
Number of babies with cerebral palsy | 18 to 22 months
  Cerebral palsy with a Gross Motor Function Classification Score >1
Number of babies with microcephaly | 18 to 22 months
  Head circumference more than 2 standard deviations below the mean
Number of babies with gastric bleeds | During neonatal hospitalisation (Expected average of 2 weeks)
  Fresh blood > 5 ml from nasogastric tube
Number of babies with persistent pulmonary hypertension | During neonatal hospitalisation (Expected average of 2 weeks)
  Severe hypoxemia disproportionate to the severity of lung disease with a significant pre-and post ductal saturation difference on pulse oximetry
Number of babies with coagulopathy | During neonatal hospitalisation (Expected average of 2 weeks)
  Prolonged blood coagulation requiring blood products
Number of babies with intracranial haemorrhage | During neonatal hospitalisation (Expected average of 2 weeks)
  Major parenchymal or intraventricular bleed on cranial ultrasound or magnetic resonance imaging.
Number of babies with culture-proven sepsis | During neonatal hospitalisation (Expected average of 2 weeks)
  Isolation of a pathogenic organism from blood or cerebrospinal fluid along with clinical evidence of sepsis or elevation of C-reactive protein
Number of babies with severe thrombocytopenia | During neonatal hospitalisation (Expected average of 2 weeks)
  Platelet count of less than 25 000 per μL or less than 50 000 per μL with active bleeding
Number of babies with abnormal neurological examination at discharge | During neonatal hospitalisation (Expected average of 2 weeks)
  Structured neurological examination as per the NICHD NRN trial (Shankaran et al NEJM 2005) discharge exam criteria

OTHER OUTCOMES:
Basal ganglia/thalami magnetic resonance (MR) Lactate/NAA peak area ratio | 10 to 14 days after birth
  Lactate/NAA peak area metabolic rations in the deep brain nuclei on proton MR spectroscopy
Basal ganglia/thalami magnetic resonance (MR) NAA/Creatine peak area ratio | 10 to 14 days after birth
  NAA/Creatine peak area metabolic rations in the deep brain nuclei on proton MR spectroscopy
White matter magnetic resonance (MR) NAA/Creatine peak area ratio | 10 to 14 days after birth
  NAA/Creatine peak area metabolic rations in the White matter on proton MR spectroscopy
White matter magnetic resonance (MR) Lactate/NAA peak area ratio | 10 to 14 days after birth
  Lactate/NAA peak area metabolic rations in the White matter on proton MR spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, PhD, Principal Investigator — Imperial College London
Locations (10):
- Bangladesh (2):
  - Bangabandhu Sheikh Mujib Medical University, Dhaka
  - Dhaka Medical College, Dhaka
- India (7):
  - Aurangabad Medical College, Aurangabad
  - Bangalore Medical College, Bangalore
  - Indira Gandhi Institute of Child Health, Bangalore
  - Institute of Child Health, Madras Medical College, Chennai
  - Kasturba Gandhi Medical College, Chennai
  - Karnataka Institute of Medical Sciences, Hubli
  - Lokmanya Tilak Municipal Medical College, Mumbai
- University of Kelaniya, Kelaniya, Sri Lanka

IPD SHARING:
Plan to Share IPD: Yes
Protocol, SAP, consent forms
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Protocol, SAP and consent forms will be shared midway through the trial recruitment following appropriate requests

REFERENCES:
- [Background] Ivain P, Montaldo P, Khan A, Elagovan R, Burgod C, Morales MM, Pant S, Thayyil S. Erythropoietin monotherapy for neuroprotection after neonatal encephalopathy in low-to-middle income countries: a systematic review and meta-analysis. J Perinatol. 2021 Sep;41(9):2134-2140. doi: 10.1038/s41372-021-01132-4. Epub 2021 Jun 26. PMID 34175900
- [Background] Thayyil S, Pant S, Montaldo P, Shukla D, Oliveira V, Ivain P, Bassett P, Swamy R, Mendoza J, Moreno-Morales M, Lally PJ, Benakappa N, Bandiya P, Shivarudhrappa I, Somanna J, Kantharajanna UB, Rajvanshi A, Krishnappa S, Joby PK, Jayaraman K, Chandramohan R, Kamalarathnam CN, Sebastian M, Tamilselvam IA, Rajendran UD, Soundrarajan R, Kumar V, Sudarsanan H, Vadakepat P, Gopalan K, Sundaram M, Seeralar A, Vinayagam P, Sajjid M, Baburaj M, Murugan KD, Sathyanathan BP, Kumaran ES, Mondkar J, Manerkar S, Joshi AR, Dewang K, Bhisikar SM, Kalamdani P, Bichkar V, Patra S, Jiwnani K, Shahidullah M, Moni SC, Jahan I, Mannan MA, Dey SK, Nahar MN, Islam MN, Shabuj KH, Rodrigo R, Sumanasena S, Abayabandara-Herath T, Chathurangika GK, Wanigasinghe J, Sujatha R, Saraswathy S, Rahul A, Radha SJ, Sarojam MK, Krishnan V, Nair MK, Devadas S, Chandriah S, Venkateswaran H, Burgod C, Chandrasekaran M, Atreja G, Muraleedharan P, Herberg JA, Kling Chong WK, Sebire NJ, Pressler R, Ramji S, Shankaran S; HELIX consortium. Hypothermia for moderate or severe neonatal encephalopathy in low-income and middle-income countries (HELIX): a randomised controlled trial in India, Sri Lanka, and Bangladesh. Lancet Glob Health. 2021 Sep;9(9):e1273-e1285. doi: 10.1016/S2214-109X(21)00264-3. Epub 2021 Aug 3. PMID 34358491
- [Derived] Garegrat R, Londhe A, Manerkar S, Fattepur S, Deshmukh L, Joshi A, Chandriah S, Kariyappa M, Devadas S, Ethirajan T, Srivasan K, Kamalarathnam C, Balachandran A, Krishnan E, Sahayaraj D, Bandiya P, Shivanna N, Burgod C, Thayyil A, Alocious A, Lanza M, Muraleedharan P, Pant S, Venkateswaran H, Morales MM, Montaldo P, Krishnan V, Kalathingal T, Joshi AR, Vare A, Patil GC, Satyanathan BP, Hapat P, Deshmukh A, Shivarudhrappa I, Annayappa MK, Baburaj M, Muradi C, Fernandes E, Thale N, Jahan I, Shahidullah M, Choudhury SM, Dey SK, Neogi SB, Banerjee R, Rameh V, Alobeidi F, Grant E, Juul SE, Wilson M, Vita E, Pressler R, Bassett P, Shankaran S, Thayyil S. Early and extended erythropoietin monotherapy after hypoxic ischaemic encephalopathy: a multicentre double-blind pilot randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2024 Oct 18;109(6):594-601. doi: 10.1136/archdischild-2024-327107. PMID 38729748